CLINICAL TRIAL: NCT01208116
Title: A Prospective Study on Predictive Value of Non-Invasive Atherosclerotic Measurements in Elderly Chinese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Sun Ning, Geriatrics Department, Tianjin Medical University General Hospital
Other Study IDs: B2009A055
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Atherosclerosis; Cardiovascular Disease
Keywords: Atherosclerosis; Prognosis; Flow-mediated dilatation; Brachial-ankle pulse wave velocity; Carotid Intimal-Medial Thickness; coronary artery calcification score; Ankle-brachial index
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subgroups: According to the demographic features, subjects may be divided into some subgroups.
  Interventions: Other: Cardiovascular events

INTERVENTIONS:
Other: Cardiovascular events — * Coronary intervention
  * Infarction
  * Congestive heart failure
  * Stroke
  * Cardiac death

SUMMARY:
The purpose of this study is to determine whether non-invasive atherosclerotic measurements (baPWV, IMT, FMD, CACS, ABI) are valuable predictors for cardiovascular events in elderly. At inception, routine physical examination and non-invasive atherosclerotic measurements will conducted on all participants. Then they will be followed prospectively for at least 2 years. All cardiovascular and other health events will be recorded.

DETAILED DESCRIPTION:
Cardiovascular disease is the most common cause of morbidity and mortality in the world, especially in elderly. Conventional risk factors are widely used in clinical practice, but it is inadequate and inaccurate due to no direct evaluation of artery. However, invasive method, it is difficult to be applied in atherosclerosis screening and only used in advanced institutions, is expensive and unacceptable. We are trying to assess the value of noninvasive measurements in predicting cardiovascular events.

Five invasive methods will be applied in the study, including

* brachial-ankle Pulse Wave Velocity(baPWV)
* Carotid Intimal-Medial Thickness(CIMT)
* Flow Mediated Dilation(FMD)
* Ankle-Brachial Index(ABI)
* Coronary Artery Calcification Score(CACS)

These indices represent not only different phase of atherosclerosis, but also various sections and arterial layers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, age>=60, no gender restriction.
* To be able to apply the measurement mentioned above.
* Medical history are maintained precisely.
* Tianjin Medical University General Hospital is the participants' designated hospital by national health authority.

Exclusion Criteria:

* Systemic inflammation.
* Malignant tumor
* Chronic lung disease
* Liver disease
* Aortic aneurysm

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with an age>=60 years, who are designated for healthcare in Tianjin Medical University General Hospital will be enrolled in the study and there is no restriction on gender. Medical histroy are recorded precisely. The protocol was approved by our Institutional Ethics Committee and all subjects give informed consent before participating.
Sampling Method: Non-Probability Sample
Enrollment: 1290 (Estimated)
Dates: Start 2010-04

CONTACTS AND LOCATIONS:
Overall Officials: Ning Sun, M.D., Study Director — Tianjin Medical University General Hospital
Locations (1):
- Geriatric Department, Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China